CLINICAL TRIAL: NCT03915405
Title: An Open-label, Phase 1 Study of KHK2455 in Combination With Avelumab in Adult Subjects With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: KHK2455 (IDO Inhibitor) Plus Avelumab in Adult Subjects With Advanced Bladder Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination was based on the business decision
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2455-002; 2018-003796-35 (EudraCT Number)
Record Dates: First submitted 2019-03-19; First posted 2019-04-16 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KHK2455 in Combination with Avelumab (Experimental)
  Interventions: Drug: KHK2455; Drug: Avelumab

INTERVENTIONS:
Drug: KHK2455 — orally, once daily.
Drug: Avelumab — IV Administration
  Other Names: Bavencio

SUMMARY:
This is a two-part (dose-escalation, dose-expansion), multicenter, open-label Phase 1 study of KHK2455 in combination with avelumab in adult subjects with locally advanced or metastatic urothelial carcinoma (including bladder, urethra, ureters, and renal pelvis).

DETAILED DESCRIPTION:
This is a two-part (dose-escalation, dose-expansion), multicenter, open-label Phase 1 study of KHK2455 in combination with avelumab in adult subjects with locally advanced or metastatic urothelial carcinoma (including bladder, urethra, ureters, and renal pelvis). Subjects will be screened for entry into this study after signing informed consent. Subjects must meet inclusion/exclusion criteria to participate in this study.

* Part 1 (dose-escalation phase) has a modified 3+3 design that will evaluate the safety and tolerability and identify the MTD or highest protocol-defined dose, in the absence of exceeding the MTD.
* Part 2 (cohort-expansion phase) will further explore the safety, pharmacokinetics, pharmacodynamics, and anti-tumor activity for the combination regimen at the MTD or highest dose level tested.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female and must be ≥ 18 years of age; have an ECOG PS of 0 or 1; and a life expectancy of > 3 months in the Investigator's judgment;
* Subjects are able to understand and willing to sign the ICF, according to institutional standards, prior to the initiation of any study related procedures
* Subjects must have histological or cytological evidence of metastatic or advanced urothelial carcinoma (including bladder, urethra, ureters, and renal pelvis that has predominantly transitional cell or urothelial features); and have measurable neoplastic disease according to RECIST v1.1 criteria
* Subjects must have been previously treated with a platinum-based therapy and progressed; OR Been previously treated with platinum based adjuvant or neo-adjuvant therapy and relapsed or progressed; OR
* Be platinum-based chemotherapy intolerant or ineligible; OR
* Have progressed during or after treatment with approved PD-1/PD-L1 inhibitors
* Subjects must have a tumor accessible for fresh biopsy at the baseline visit and for IDO assessment. If current circumstances prohibit the biopsy procedure (e.g., temporary hospital protocol restrictions, regulatory or local authority requirements, etc.) then archived tissue from previous biopsies (fresh frozen tissue < 9 months and formalin fixed-paraffin embedded [FFPE] block of ≤ 24 months) without intervening checkpoint inhibitors can substitute for a fresh baseline biopsy;
* Subjects must be able to swallow the solid (encapsulated) dosage form of KHK2455

Exclusion Criteria:

* Subjects who have been previously treated with avelumab or any IDO1 inhibitor or CTLA-4, PD-1/PD-L1 checkpoint inhibitors; or any investigational immunotherapy including but not limited to anti-cancer vaccines or oncotropic viruses
* Subjects with prior or current liver metastases;
* Subjects with a history of organ transplant or allogeneic bone marrow transplant;
* Subjects with pre-existing uveitis or other known clinically meaningful retinal disorders as determined by a local ophthalmologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | up to 24 months
  To characterize the safety and tolerability of KHK2455 administered in combination with avelumab in subjects with locally advanced or metastatic urothelial carcinoma (including bladder, urethra, ureters, and renal pelvis).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Kyowa Research Site USA001, St. Petersburg, Florida
  - Kyowa Research Site USA005, Iowa City, Iowa
  - Kyowa Research Site USA006, Santa Fe, New Mexico
  - Kyowa Research Site USA 009, Houston, Texas
  - Kyowa Research Site USA007, Milwaukee, Wisconsin
- Spain (4):
  - Kyowa Research Site ESP002, Barcelona
  - Kyowa Research Site ESP003, Barcelona
  - Kyowa Research Site ESP004, Madrid
  - Kyowa Research Site ESP001, Madrid